CLINICAL TRIAL: NCT05976282
Title: Addressing Colorectal Cancer in South Florida Firefighters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Florida (Other)
Responsible Party: Principal Investigator, Erin Kobetz-Kerman, PhD, MPH, Professor, University of Miami
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 20150905; NCI-2023-00172 (Registry Identifier: NCI Clinical Trials Reporting Program (NCI CTRP))
Record Dates: First submitted 2023-07-27; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07

CONDITIONS: Colorectal Cancer; CRC
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FIT Group (Experimental): Participants aged 40-65 years will receive the self-administered FIT test by mail including instructions for obtaining and returning their stool specimens. Participants will be in this group for up to 6 months.
  Interventions: Other: Fecal Immunochemical Test
- Septin9 Test Group (Experimental): Participants aged 50-65 years who declined the initial offer of FIT, will complete a 10-15 minute questionnaire about their personal health, quality of life, and health-related to colorectal cancer including screening history and smoking. Participants will be in this group for up to 6 months.
  Interventions: Other: Septin9 Test

INTERVENTIONS:
Other: Fecal Immunochemical Test — The Fecal Immunochemical Test (FIT) is self-administered one-time for participants, per standard of care. This allows participants to obtain their own stool specimens from bowel movements without having a regular colorectal screening procedure in the doctor's office. Participants will use the FIT at the time of their next bowel movement and return their specimens to the laboratory by mail on the same or next day.
  Other Names: FIT
  Arms: FIT Group
Other: Septin9 Test — Septin9 (SEPT9) is a blood-based test that will be offered to eligible participants one-time who refused the FIT. Participants will undergo a blood draw collected by a nurse or certified phlebotomist, 90 days after their refusal of the initial offer of FIT.
  Other Names: SEPT9
  Arms: Septin9 Test Group

SUMMARY:
The standard way of screening for colorectal cancer is to have a series of fecal blood tests, where a sample is taken from a participant's stool, or an endoscopic procedure performed by a doctor, where a camera is used to look inside the bowel. This research study will use a test performed by the participant. This test will look for changes in the stool that can identify if participants are at higher risk for cancer.

Another aim of this study is to better understand what firefighters and retired firefighters think about colorectal cancer and other health issues. This information will help us develop programs that may improve colorectal cancer outcomes in the firefighter community.

ELIGIBILITY:
Inclusion Criteria:

* For this study, participation is open to active and retired firefighters:

  1. ≥ 40 and ≤ 65 years of age,
  2. who work or worked in Florida Fire and Rescue departments and
  3. report never having fecal occult blood test (FOBT) or sigmoidoscopy/colonoscopy in their life or only one FOBT in the past year, a sigmoidoscopy in the last 5 years or a colonoscopy in the last 10 years. The research assistant will assess eligibility using a brief screener that will be completed online via RedCAP.
* For years 2 and 3 of the study, the investigators will enroll previously eligible participants who did not complete colorectal cancer (CRC) screening during year 1. The investigators will also enroll participants who completed fecal immunochemical test (FIT) with our study during year 1 and 2. They will be contacted via RedCAP and a follow up phone call at the 1 year mark of their previous screening. Based on national guidelines, FIT screening is suggested on a yearly basis. The eligibility criteria will be the same and participants will sign a revised informed consent form, stating that they understand that they are being re-consented for the same study.
* Participants, ages 50-65 years old, meeting the above criteria who declined the offered standard-of-care FIT will then be offered the blood-based septin9 test 90 days from the initial offering. FDA guidelines require the participant to be at least 50 years old to participate in the septin9 blood collection. The blood based test will be collected by a nurse or certified phlebotomist in the community setting.

Exclusion Criteria:

* Individuals, who have a personal history of CRC, inflammatory bowel disease (ie, Crohn disease involving the colon or ulcerative colitis) will be excluded from participation as these conditions increase the likelihood of positive test results not associated with the onset or recurrence of CRC disease. Additionally, individuals will be excluded if they are not physically capable of performing the FIT themselves.
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 646 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2019-11-19 (Actual)

PRIMARY OUTCOMES:
Feasibility of Participants Completing FIT Screening Tool | Up to 6 months
  Feasibility will be measured as the percentage of eligible participants completing the FIT screening tool. Criterion for success: 65% of all eligible participants complete the FIT screening tool.
Feasibility of FIT Specimens Adequate for Lab Processing | Up to 6 months
  Feasibility will be measured as the percentage of FIT specimens collected from participants that are adequate for processing. Criterion for success: 95% of all FIT specimens are adequate for lab processing.
Feasibility of Participants with Positive FIT Results Who Comply with Follow-up for Colonoscopy | Up to 6 months
  Feasibility will be measured as the percentage of participants with positive FIT results who comply with the necessary follow-up for colonoscopy. Criterion for success: 85% of all participants with positive FIT results comply with necessary follow up for colonoscopy.
Acceptability of Participants Who Feel FIT is an Acceptable Method of Screening | Up to 6 months
  Acceptability will be measured as the percentage of participants who feel the FIT is an acceptable method of screening. Criterion for success: 90% of participants who complete the FIT find it to be an acceptable method of screening.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Kobetz-Kerman, Phd, MPH, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No